CLINICAL TRIAL: NCT06720220
Title: Sedation Using Dexmedetomidine With or Without Different Methods of Airway Topical Anesthesia for Awake Fiberoptic Nasal Intubation in Patients Undergoing Elective Surgeries Under General Anesthesia
Brief Title: Role of Airway Topicalization in Awake Fiberoptic Intubation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Airway topicalization
Record Dates: First submitted 2024-07-11; First posted 2024-12-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2024-12

CONDITIONS: Airway Complication of Anesthesia
Keywords: Dexmedetomidine, Airway Topicalization, AFOI
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group C (Sedation / Control group) (Placebo Comparator): The patients will receive only dexmedetomidine as a sedative for AFOI with placebo airway topicalization by nebulization, atomization and spray as you go using normal saline 0.9%.
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Group N (Nebulization group) (Active Comparator): The patients will receive dexmedetomidine as a sedative in addition to lidocaine 2% nebulization for airway topicalization and placebo airway topicalization by atomization and "spray as you go" using normal saline 0.9%.
  Interventions: Drug: Dexmedetomidine Hydrochloride; Other: Nebulization
- Group A (Atomization group) (Active Comparator): The patients will receive dexmedetomidine as a sedative in addition to lidocaine 2% by atomization "modified McKenzie technique" and placebo airway topicalization by nebulization and "spray as you go" using normal saline 0.9%.
  Interventions: Drug: Dexmedetomidine Hydrochloride; Other: Atomization
- Group S (SAYGo group) (Active Comparator): The patients will receive dexmedetomidine as a sedative in addition to lidocaine 2% by "Spray as You Go" technique and placebo airway topicalization by atomization and nebulization using normal saline 0.9%.
  Interventions: Drug: Dexmedetomidine Hydrochloride; Other: Spray-As-You-Go

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — procedural sedation by I.V. infusion of dexmedetomidine. It was prepared as 200 ug (2 ml) of dexmedetomidine added to 48 ml of 0.9% saline.
  A loading dose of dexmedetomidine 0.5 to 1 ug/kg was given over 10- 20 minutes, followed by 0.2-0.7 ug/kg/hr as a continuous infusion by a syringe pump. During the dexmedetomidine infusion, a spontaneous respiratory pattern was maintained, and the level of sedation achieved to a point of semi-sleep but responds to commands (equivalent to Modified Ramsay Sedation Scale score of 3).
  Other Names: Precedex
Other: Nebulization — nebulization session through a face mask nebulizer attached to an oxygen source. The nebulizer chamber was filled with 10 ml of 2% lidocaine (200 mg). The oxygen flow was adjusted at a rate of 8-10 L/min for 10-15 minutes.
  Arms: Group N (Nebulization group)
Other: Atomization — Airway topicalization by atomization (through a modification of McKenzie technique). This modification utilizes a 10-Fr suction catheter instead of 20-gauge cannula. This suction catheter was attached to oxygen tubing with a three-way stopcock. The oxygen tubing was attached to an oxygen source, which delivers a flow of 2-4 L/min. A 10-ml syringe filled with 10 ml of lidocaine 2% was attached to top port of the three-way stopcock.
  Local anesthetic was injected via the syringe forming a jet- like spray for topicalization of the nasal and oral mucosa
  Arms: Group A (Atomization group)
Other: Spray-As-You-Go — airway topicalization method using the fiberoptic bronchoscope itself. The fiberoptic bronchoscope, preloaded with a 6.5 or 7 mm endotracheal tube, was passed under direct vision through the nose into the pharynx. Then 10-ml syringe containing 10 ml Lidocaine 2%, was attached to the working channel, and thus the local anesthetic was sprayed towards the mucosa of postnasal space and back of throat, while advancing the fiberscope. At the level of the epiglottis and around the vocal cords 2-4 ml of lidocaine 2% were sprayed toward these structures as the patient takes a deep breath to achieve sufficient anesthesia to the laryngeal inlet. The patient was asked to take another deep breath as the scope was passed through the vocal cords and 2 ml of lidocaine 2% is sprayed to the trachea and the scope was advanced further until the carina was visualized.
  Arms: Group S (SAYGo group)

SUMMARY:
Airway management is an integral part of general anesthesia. Difficult airway management may lead to various adverse events such as airway trauma, up to cardiopulmonary arrest.

Awake fiberoptic intubation is the gold standard technique for difficult airway, although it can lead to significant patient anxiety and discomfort. Thus, it necessitates sufficient airway anesthesia for the patient's comfort and cooperation.

One challenge associated with this procedure is providing adequate anxiolysis while maintaining a patent airway and adequate ventilation. Suppressing airway reflexes represents another challenge to achieve successful airway management.

Sedation can be used during such procedures for better patient cooperation. The ideal sedative for awake intubation would provide patient comfort and good intubating conditions and at the same time maintain a patent airway.

Dexmedetomidine is a selective alpha-2-adrenoceptor agonist that can cause sedation, anxiolysis, sparing with minimal respiratory depression. It reduces the salivary secretion, which is advantageous for awake fiberoptic intubation.

Airway nerve blocks are considered technically difficult to perform and generally carry a higher risk of complications, including bleeding, nerve damage, and intravascular injection, but if performed by an experienced anesthesiologist, they would achieve excellent airway anesthesia for successful AFOI.

There are various airway topical techniques such as nebulization, atomization (McKenzie technique), and Spray-As-You- Go technique.

In the present study, we try to find out which is more effective for topicalization to achieve good intubating conditions in patients undergoing awake fiberoptic nasotracheal intubation using different methods of airway topicalization, nebulization, atomization or We used a modification of the McKenzie technique for atomization.

DETAILED DESCRIPTION:
-Type of the Study: Prospective randomized double-blind controlled clinical trial.

- Randomization: 56 patients were included in this prospective randomized double-blind controlled clinical study. They were randomized by computer-generated randomization table into 4 equal groups (14 patients each):

* Group C (Sedation / Control group) (n=14) patients received only dexmedetomidine as a sedative with placebo airway topicalization by nebulization, atomization, and spray as you go using normal saline 0.9%.
* Group N (Nebulization group) (n=14) patients received dexmedetomidine as a sedative in addition to lidocaine 2% nebulization for airway topicalization and placebo airway topicalization by atomization and spray as you go using normal saline 0.9%.
* Group A (Atomization group) (n=14) patients received dexmedetomidine as a sedative in addition to lidocaine 2% by atomization "modified McKenzie technique" and placebo airway topicalization by nebulization and spray as you go using normal saline 0.9%.
* Group S (SAYGo group) (n=14) patients received dexmedetomidine as a sedative in addition to lidocaine 2% by "Spray As You Go" technique and placebo airway topicalization by atomization and nebulization using normal saline 0.9%.

A well-trained nurse prepared different topicalization methods according to each group. The anesthesiologist who performed the awake fiberoptic nasal intubation and followed the perioperative data was unaware of each preparation, as well as the patient to ensure blindness of the study.

- Preoperative Preparation:

The day before surgery, all participating patients were interviewed, the procedure of awake fiberoptic intubation was explained and a written informed consent was obtained from each patient. General and airway examination was done to rule out any contraindication. All patients were investigated by complete blood count, liver function tests, kidney function tests, and coagulation profile. All patients were kept fasting for minimum of 2 hours for clear liquids and 6 hours for solid food before the operation.

On the day of surgery, in the pre-anesthesia room, two 20-gauge cannulae were inserted, secured and maintenance intravenous fluid (ringer lactate) infusion was started via one of them while the other for continuous infusion of sedative drug.

Premedication was done with atropine 1 mg I.M. and metoclopramide 10 mg I.V. 1 hour before conducting the technique. Xylometazoline hydrochloride decongestant nasal drops and lignocaine gel 2% were applied in both nasal passages. A gauze soaked in 10 ml lidocaine 2% was placed in the oral cavity for 10 minutes.

- Intraoperative:

On arrival to the operating room, standard monitoring including non-invasive blood pressure, electrocardiogram, and pulse oximetry was performed on all patients. Baseline readings of mean arterial pressure, heart rate, and oxygen saturation were recorded. Supplemental oxygen was administered at 6-8 L/min via nasal prongs through patient's mouth.

Sedation technique:

All patients in all groups received procedural sedation by I.V. infusion of dexmedetomidine. It was prepared as 200 µg (2 ml) of dexmedetomidine added to 48 ml of 0.9% saline. A loading dose of dexmedetomidine 0.5 to 1 µg/kg was given over 10- 20 minutes, followed by 0.2-0.7 µg/kg/hr as a continuous infusion by a syringe pump. During the dexmedetomidine infusion, a spontaneous respiratory pattern was maintained, and the level of sedation achieved to a point of semi-sleep but response to commands (equivalent to a Modified Ramsay Sedation Scale score of 3). The total dose of dexmedetomidine used to reach this point of sedation in each group was calculated and recorded.

Nebulization Technique:

Patients in the nebulization group received procedural sedation by I.V. infusion of dexmedetomidine as mentioned before, then they had a nebulization session through a face mask nebulizer attached to an oxygen source. The nebulizer chamber was filled with 10 ml of 2% lidocaine (200 mg). The oxygen flow was adjusted at a rate of 8-10 L/min for 10-15 minutes. (200 mg of which 25% is typically absorbed = 50 mg) into the nasopharynx & oropharynx.

The patient was asked to take shallow breaths to topicalize the more proximal airway and to take slow deep breaths for the more distal airway. This process may need repeating to ensure adequate airway anesthesia. Adequate topical anesthesia was confirmed by heaviness or numbness of the tongue.

To rule out bias, nebulization was done using 10 ml of normal saline 0.9% to patients in other groups.

Atomization technique:

Patients in the atomization group received procedural sedation by I.V. infusion of dexmedetomidine as mentioned before, then they were subjected to airway topicalization by atomization (through a modification of the McKenzie technique). This modification utilizes a suction catheter instead of a 20-gauge cannula (to allow the local anesthetic drug to topicalize the more distal airway creating a jet-like spray of local anesthetic towards airway mucosa). This suction catheter was attached to oxygen tubing with a three-way stopcock. The oxygen tubing was attached to an oxygen source, which delivers a flow of 2-4 L/min. A 10-ml syringe filled with 10 ml of lidocaine 2% was attached to the top port of the three-way stopcock

As the local anesthetic was administered via the syringe, a jet-like spray was created to enable effective topicalization of the nasal and oral mucosa. The spray should be targeted to the nasal passage, soft palate, uvula, base of tongue and posterior pharyngeal wall. The patient was asked to spit out or swallow the local anesthetic after gargling. Once swallowed it is removed by liver following first pass metabolism without adverse effects.

To rule out bias, atomization was done using 10 ml normal saline 0.9% to patients in other groups.

Spray as you go (SAYGo) Technique:

Patients in the SAYGo group received procedural sedation by I.V. infusion of dexmedetomidine as mentioned before, then they were subjected to airway topicalization method using the fiberoptic bronchoscope itself. The fiberoptic bronchoscope, preloaded with a 6.5 or 7 mm endotracheal tube, was passed under direct vision through the nose and into the pharynx. Then 10-ml syringe containing 10 ml Lidocaine 2%, was attached directly to the working channel, and thus the local anesthetic was sprayed to target the mucosa of the postnasal space and back of the throat, as the fiberscope was advanced through the airway.

At the level of the epiglottis and around the vocal cords 2-4 ml of lidocaine 2% were sprayed toward these structures as the patient takes a deep breath to achieve sufficient anesthesia to the laryngeal inlet. The patients are informed that they may cough. If the patient coughs, it is prudent to wait until the view clears.

The patient was asked to take another deep breath as the scope was passed through the vocal cords and 2 ml of lidocaine 2% is sprayed to the trachea and the scope was advanced further until the carina was visualized.

Awake Nasotracheal Fiberoptic Intubation Technique:

After the patient prepared with sedation either alone or with airway topicalization, the patient's head was positioned neutrally or slightly extended. The Fiberoptic Bronchoscope preloaded with an appropriate size endotracheal tube (size 7.0 mm internal diameter for male patients and size 6.5 mm for female patients) was lubricated with water-soluble gel to decrease friction and facilitate insertion. The tip of the fiberoptic bronchoscope was inserted into the more patent nostril and advanced through the nasal passage, entering the pharynx, then the tip of the scope was deflected upward till the epiglottis was seen in the midline. The scope was advanced beneath the epiglottis till the vocal cords were visualized. The patient was asked to take a deep breath so the scope could pass between the vocal cords observing the tracheal rings and reaching the carina. Then the patient was asked to take a deep breath, the lubricated endotracheal tube "preloaded on the scope" at the entrance to the nose is rotated through the nose and into the trachea along the fiberoptic bronchoscope. The patient was informed that this may be uncomfortable.

Once the tube had successfully been passed into the trachea, its depth was noted, verifying that the tube is in the trachea by observing the carina and the scope was finally removed.

In all groups, once the tube position was confirmed (using a stethoscope and capnography), the patient was anesthetized using propofol 2 mg/kg i.v, rocuronium 0.6-0.9 mg/kg i.v and the cuff of the endotracheal tube was inflated. Anesthesia was maintained with inhalation of oxygen and isoflurane 1.5% minimal alveolar concentration (MAC), rocuronium 0.15 mg/kg i.v increments and the surgical procedure was proceeded as planned.

Patients' intubation condition was assessed by:

1. Five-point fiberoptic intubation comfort score during bronchoscopy as follows: (0: no reaction, 1: slight grimacing, 2: heavy grimacing, 3: verbal objection, 4: defensive movements).
2. patients' behavior was assessed using three-point behavior score immediately after intubation as follows: (0: cooperative, 1: restless/minimal resistance, 2: severe resistance).
3. Bronchoscopy-guided intubation time (from the insertion of the fiberoptic bronchoscope in the nostril to confirmation of tracheal intubation by capnography).

Vital parameters (MAP, HR) and oxygen saturation (SpO2%) were continuously monitored & recorded immediately after intubation, every 5 min during the 1st 15 min then every 15 min till 1 hour. Any changes in MAP, HR or any hypoxic episode (SpO2 <90%) during intubation were recorded.

Four-point patient satisfaction score (0: excellent, 1: good, 2: reasonable, 3: poor) was used to assess patient satisfaction post-operatively.

Postoperative adverse events such as sore throat, hoarseness or any signs of lidocaine toxicity such as ECG changes, seizures, and bronchoconstriction were noted.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance and willingness to sign a written informed consent document.
* Body mass index (BMI): 18.5 - 24.9 kg/m2.
* American Society of Anesthesiologists physical status: class I & II.
* patients undergoing elective surgery under general anesthesia.

Exclusion Criteria:

* Patient refusal.
* Patients with known allergies to study drugs.
* Patients having any contraindication to nasal intubation; nasal bleeding or infection.
* Patients having bleeding disorders.
* Reactive airway disease.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Assessment of patients' intubation condition during awake fiberoptic intubation. | 1 - 3 hours
  The patients' intubation condition is assessed by the Five-point fiberoptic intubation comfort score

SECONDARY OUTCOMES:
Calculation of the total dexmedetomidine dose used for sedation | 20 minutes
  the total dexmedetomidine dose used during the procedure
Peri-intubation measurement of mean arterial pressure . | 1 hour
  measurement of the mean arterial pressure every 2 minutes for the first hour.
Peri-intubation measurement of heart rate. | 1 hour
  measurement of the heart rate every 2 minutes for the first hour.
Evaluation the post-operative patient satisfaction | 1 hour
  Evaluating the post-operative patient satisfaction by the Four-point patient satisfaction Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Howaida Kamal Abdellatif, MD, Study Director — Professor of Anesthesia, Intensive Care and pain management
Locations (1):
- Faculty of medicine - Zagazig University, Zagazig, Alsharkia, Egypt

IPD SHARING:
Plan to Share IPD: No